CLINICAL TRIAL: NCT06330402
Title: Undersøgelse af sammenhængen Mellem Biomekanik og Smerter Ved Gang
Brief Title: Exploration of Gait Biomechanics and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristian Kjær Petersen (Other)
Responsible Party: Sponsor-Investigator, Kristian Kjær Petersen, Principal Investigator, Aalborg University
Organization: Aalborg University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20220063
Record Dates: First submitted 2024-03-12; First posted 2024-03-26 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Pain; Healthy
MeSH Terms: conditions — Pain | interventions — Saline Solution, Hypertonic; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Painful condition (Experimental): Hypertonic saline injection to the infrapatellar fat pad.
  Interventions: Other: Hypertonic saline injection
- Control condition (Placebo Comparator): Isotonic saline injection to the infrapatellar fat pad.
  Interventions: Other: Isotonic saline injection

INTERVENTIONS:
Other: Hypertonic saline injection — 0.25 mL injection with hypertonic saline (7%) to the infrapatellar fat pad.
  Arms: Painful condition
Other: Isotonic saline injection — Control injection with 0.25 mL isotonic saline (0.9%) to the infrapatellar fat pad.
  Arms: Control condition

SUMMARY:
This interventional study aims to test gait biomechanics in healthy individuals with and without experimental knee pain. The main questions it aims to answer are:

* How do gait patterns change during painful walking?
* Can pain sensitivity testing and gait biomechanics predict experimental knee pain intensity?

Participants will receive two knee injections: a) Hypertonic saline (painful condition) and b) Isotonic saline (control condition).

DETAILED DESCRIPTION:
This study will be a randomized, crossover design where experimental knee pain will be provoked in healthy subjects using hypertonic saline injections to the infrapatellar fat pad (IFP). This will be controlled with a second injection of isotonic saline, which is non-painful. The participants will not be informed of the type of injection.

Hypertonic saline injections to the IFP usually provoke pain lasting about 15 minutes. Within this timeframe, motion capture will be conducted to estimate the biomechanics of gait. During the motion capture the participants will perform five 10-meter walking trials and three jumps. This process will be replicated for the control condition.

Additionally, the participants will have their pain sensitivity tested using cuff-pressure algometry before both IFP injections.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged 18-45 years

Exclusion Criteria:

* Pregnancy
* Drug addiction, defined as the use of cannabis, opioids, or other drugs
* Previous or current neurologic or musculoskeletal illnesses
* Current pain
* Lack of ability to cooperate

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Infrared marker XYZ coordinates | Baseline
  Marker-based motion capture with infrared cameras will be used to estimate placement of reflective markers in the XYZ planes measured in milimeters. Reflective markers will be placed from head-to-toe on anatomical landmarks.
Pain sensitivity. | Baseline
  Cuff-pressure algometry will be used to estimate pressure detection and tolerance thresholds, temporal summation of pain, and conditioned pain modulation.

SECONDARY OUTCOMES:
The Pittsburgh Sleep Quality Index score | Baseline
  19 items summarized to a single score ranging from zero to 21 with higher scores reflecting worse quality of sleep.
The Pain catastrophizing Scale score | Baseline
  13 items summarized to a single score ranging from zero to 52 with higher scores reflecting more catastrophizing.
The Hospital Anxiety and Depression Scale | Baseline
  14 items summarized into two 7-item subscales measuring symptoms of anxiety and depression. Each subscale score ranges from zero to 21 with higher scores reflecting more severe symptoms.
Knee symptoms | Baseline
  42 items divided into five subscales: pain (9 items), activities of daily living (17 items), sport and recreation function (5 items), knee-related quality of life (4 items), and other symptoms (7 items). Each subscale is score from zero to 100 with higher scores reflecting increased severity of knee problems.
Ground reaction forces | Baseline
  Ground reaction forces will be measured in Newton-meters with force plates embedded in the floor.
Ground reaction moments | Baseline
  Ground reaction moments will be measured in Newton-meters with force plates embedded in the floor.
Ground contact XZ location | Baseline
  Ground contact XZ coordinate location will be measured in milimeters with force plates embedded in the floor.
Muscle activation | Baseline
  Muscle activation will be measured in micro-volts using wireless EMG on the muscles of the lower extremities.

OTHER OUTCOMES:
Pain intensity (NRS 0-10) | Baseline
  Pain during intervention is measured continuously every 30 seconds on a numeric rating scale from 0 'no pain' to 10 'the worst pain imagineable'
Pain distribution | Baseline
  Pain during intervention is marked on a body chart

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided